CLINICAL TRIAL: NCT00823836
Title: Clinical Evaluation of Ropinirole PR/XR Tablet for Adjunctive Therapy to L-dopa in Subjects With Advanced Parkinson's Disease
Brief Title: Clinical Evaluation of Ropinirole Prolonged Release/Extended Release (PR/XR) Tablet for Adjunctive Therapy to L-dopa in Subjects With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106066
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2011-10-07 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson Disease
Keywords: Ropinirole, advanced Parkinson's disease, L-dopa adjunctive therapy
MeSH Terms: conditions — Parkinson Disease | interventions — ropinirole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropinirolePR-PR group (Experimental)
  Interventions: Drug: ropinirole PR/XR
- ropiniroleIR-PR group (Active Comparator)
  Interventions: Drug: ropinirole PR/XR; Drug: ropinirole IR

INTERVENTIONS:
Drug: ropinirole PR/XR — Double-blind non-inferiority verification phase (24 weeks) At the baseline visit (Week 0), subjects who completed screening period will be randomised (1:1) to double-blind treatment with either ropinirole PR-PR group or ropinirole IR-PR group.
  The subjects'dose will be titrated according to the recommended schedule to achieve an optimal therapeutic response (ropinirolePR/XR2-15 mg/day ,ropinirolIR0.75-15 mg/day).
  Double-blind PR/XR switching phase (8 weeks) Ropinirole IR-PR subjects will be switched overnight to a similar dose of ropinirole PR/XR, while the remaining ropinirole PR-PR group will continue on the same dosage.
  Double blind long-term treatment phase (22 weeks) The same dose level at the end of PR/XR switching phase will be continued till week 54 under blind.
  Down titration phase Subjects who complete Week 54 or withdrawn will be down titrated over a 1 to 4 weeks period.
  Other Names: ropinirole IR-PR group
Drug: ropinirole IR — Double-blind non-inferiority verification phase (24 weeks) At the baseline visit (Week 0), subjects who completed screening period will be randomised (1:1) to double-blind treatment with either ropinirole PR-PR group or ropinirole IR-PR group.
  The subjects'dose will be titrated according to the recommended schedule to achieve an optimal therapeutic response (ropinirolePR/XR2-15 mg/day ,ropinirolIR0.75-15 mg/day).
  Double-blind PR/XR switching phase (8 weeks) Ropinirole IR-PR subjects will be switched overnight to a similar dose of ropinirole PR/XR, while the remaining ropinirole PR-PR group will continue on the same dosage.
  Double blind long-term treatment phase (22 weeks) The same dose level at the end of PR/XR switching phase will be continued till week 54 under blind.
  Down titration phase Subjects who complete Week 54 or withdrawn will be down titrated over a 1 to 4 weeks period.
  Arms: ropiniroleIR-PR group

SUMMARY:
To investigate the efficacy and the safety of ropinirole PR/XR tablets to ropinirole immediate release (IR) tablets with advanced Parkinson's disease in conjunction with L-dopa in a double-blind, parallel group comparison study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at the start of the screening

* Patients who are diagnosed with advanced Parkinson's disease (PD) with severity of the modified Hoehn & Yahr criteria Stages II-IV.
* Subjects receiving a stable dose of L-dopa for at least 4 weeks prior to screening phase and demonstrating lack of control with L-dopa therapy in the following circumstances. Wearing-off phenomena. On-off fluctuations. Delayed-on/No on phenomena. Not adequately controlled on L-dopa
* QTc<450 millisecond (msec) or <480msec for patients with Bundle Branch Block - values based on either single ECG values or triplicate electrocardiogram (ECG) averaged QTc values obtained over a brief recording period.
* Age:20 years or older(at the time of informed written consent)
* Informed consent: Patients who are able to give informed written consent in person. (i.e. patients who are capable of giving informed written consent on one's own)
* Sex: either sex. Female of child-bearing potential will be eligible for inclusion in this study. However they have to have a negative pregnancy test at the screening visit, agree to further pregnancy testing at the time points determined in study assessments and procedures and practice one of the following methods of contraception from the screening visit until the end of the follow-up examination. Abstinence. Injectable progestogen. Implants of levonorgestrel. Estrogenic vaginal ring. Percutaneous contraceptive patches. Intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label. Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. Double barrier method: condom or occlusive cap (diaphragm or cervical / vault caps) plus spermicidal agent (foam /gel / film / cream / suppository)
* Both inpatient and outpatient status.

Inclusion Criteria at the start of the non-inferiority verification phase

-Patients whose Unified Parkinson's Disease Rating Scale (UPDRS) PartIII total (on) scores is 10 points or more at week 0.

Exclusion Criteria:

* Late stage advanced subjects demonstrating incapacitating peak dose or biphasic dyskinesia on their stable dose of L-dopa.
* Patients who present serious physical signs and symptoms other than those of the PD (e.g. cardiac/hepatic/renal disorder and haematopoietic disorder). The severity refers to Grade 3 according to "the Classification of the Severity of Adverse Experiences (Pharmaceutical affairs bureau/Safety division (PAB/SD) Notification No. 80, dated 29 June 1992).
* Patients with symptomatic postural hypotension. (e.g. dizziness and syncope).
* Patients with a current or history of drug abuse or alcoholism.
* Patients who have received surgical treatment for PD in the past (e.g. pallidectomy, deep brain stimulation).
* Female patients who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study or within 30 days after the last dose of the study drug.
* Patients with chronic hepatitis typeB and/or type C which is positive of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibody.
* Patients with a history of drug allergy to ropinirole hydrochloride (HCl).
* Patients with a current or history of cancer or malignant tumor.
* Others whom the investigator (subinvestigator) considers ineligible for the study.

Exclusion criteria at the start of the non-inferiority verification phase

* Patients with severe dementia (e.g. score 3 or 4 of the UPDRS item 1 (Intellectual Impairment))
* Patients with current or history of major psychosis (e.g. schizophrenia or psychotic depression) core 3 or 4 of the UPDRS item 2 (thought disorder) or item 3(depression).
* Patients who have used any dopamine agonist within 4 weeks prior to the non-inferiority verification phase
* Patients who have been treated with the following drugs at 4 weeks or earlier before the start of the non-inferiority verification phase, and whose treatment regimen of the drug has been changed. Anticholinergic agents: trihexyphenidyl hydrochloride (e.g. Artane®), piroheptine hydrochloride (Trimol®), mazaticol hydrochloride (Pentona®), metixene hydrochloride (Cholinfall®), biperiden hydrochloride (Akineton®), profenamine (Parkin®), amantadine hydrochloride (e.g. Symmetrel®),droxidopa (Dops®), citicoline (e.g. Nicholin®), selegiline hydrochloride (FP®), entacapone, (comutan®) zonisamide, Estrogens: e.g. estriol (e.g. Estriel®), CYP1A2 inhibitors: Ciprofloxacin HCl (e.g. Ciproxan®, enoxacin and fluvoxamine).
* Patients who have been treated with any other investigational drug within 12 weeks prior to the treatment phase.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- Japan (22):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Akita
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shiga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 106066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 157 participants who were enrolled in the Non-Inferiority Verification (NV) Phase entered into the Long-term Phase after completing the Prolonged Release/Extended Release (PR/XR) Switching Phase according to the study design. The remaining participants entered into the Down-titration Phase after completing the PR/XR Switching Phase.
Groups:
- Ropinirole PR-Ropinirole PR: Participants received ropinirole prolonged release/extended release (PR/XR) tablets orally once daily. Participants firstly received matching PR/XR placebo tablets for 2 weeks and then received 2 milligram (mg) PR/XR tablets with a weekly dose increase to 4 mg at Week 4. Between Weeks 6 and 24, the dose was optionally increased at intervals of 2 weeks or longer up to 16 mg/day. In the PR/XR Switching Phase, administration of the PR/XR tablets was continued until Week 32 at the same dose level as that at the end of the Non-Inferiority Verification Phase. Participants who entered into the Long-term Phase continued to receive ropinirole PR/XR tablets until Week 54 at the same dose level as that at the end of the PR/XR Switching Phase. Participants who did not enter the Long-term Phase entered the Down-titration Phase after completion of the PR/XR Switching Phase.
- Ropinirole IR-Ropinirole PR: Participants received ropinirole immediate release (IR) tablets three times daily at the initial dose of 0.75 mg/day with a weekly dose increase to 3 mg/day at Week 4. Between Weeks 6 and 24, the dose was optionally increased at intervals of 2 weeks or longer up to 15 mg/day. Ropinirole IR tablets were administered until the night of the Week 24 visit and were replaced by ropinirole PR/XR tablets on the following morning, the morning of the first day of the PR/XR Switching Phase, at the same dose level. Participants who entered the Long-term Phase continued to receive ropinirole PR/XR until Week 54 at the same dose level as that at the end of the PR/XR Switching Phase. Participants who did not enter into the Long-term Phase entered the Down-titration Phase after completion of the PR/XR Switching Phase.
Period: NV and PR/XR Switching Phases
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Started | 156 | 146
Completed | 124 | 117
Not Completed | 32 | 29
Not completed — Adverse Event | 22 | 21
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 5 | 2
Not completed — Withdrawal by Subject | 4 | 5
Period: Long-term Phase
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Started | 73 | 84
Completed | 68 | 79
Not Completed | 5 | 5
Not completed — Adverse Event | 3 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR | Total
Number analyzed (Participants) | 156 | 146 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (7.95) | 68.3 (8.22) | 68.8 (8.08)
Gender [Count of Participants; unit: Participants]
  Female | 93 | 81 | 174
  Male | 63 | 65 | 128
Race/Ethnicity, Customized [Number; unit: participants] | 156 | 146 | 302

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Week 0 (Baseline) in the Japanese Unified Parkinson's Disease Rating Scale (UPDRS) Part III Total Score at the Final Assessment Point (FAP) (up to Week 24) in the Non-Inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of Parkinson's Disease (PD) patients objectively. Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. Mean change from Week 0 was calculated as the total score at FAP minus the total score at Week 0. Participants who withdrew before Week 2 and who had only one observation for the part III total score were not included in the analysis.
Time Frame: Week 0 and FAP (up to Week 24)
Population: Per Protocol Set (PPS): participants with exclusion from the Full Analysis Set (FAS) of those violating the study protocol and assessed to be excluded from the assessment of drug efficacy. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 141 | 133
scores on a scale | -10.8 (8.32) | -11.0 (7.56)
Statistical Analysis 1: Comparison: Ropinirole PR-Ropinirole PR vs Ropinirole IR-Ropinirole PR; Test type: Non-Inferiority or Equivalence — Non-inferiority of ropinirole PR/XR tablets to ropinirole IR tablets was assessed with a non-inferiority margin of 2.5; p = 0.702, ANCOVA — Analysis of covariance (ANCOVA) model: value of change from Week 0 at Week 24 = treatment group + Week 0 value; Median Difference (Net) = 0.34, 95% CI 2-sided [-1.41 to 2.09]

2. Secondary Outcome: Percentage of Responders on the Japanese UPDRS Part III Total Score at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: Thirty percent responders were defined as participants with a 30 percent or greater reduction from Week 0 in the Japanese UPDRS Part III total score. Twenty percent responders were defined as participants with a 20 percent or greater reduction from Week 0 in the Japanese UPDRS Part III total score. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 and who had only one measurement for the part III total score were not included in the analysis.
Time Frame: FAP (up to Week 24)
Population: FAS: participants who were progressed to the Non-Inferiority Verification Phase but excluding those who did not have the target indication, those who had not received at least one dose of investigational product, and those whose measured data in efficacy were not available after treatment initiation.
Measure: Number; unit: percentage of participants
Groups:
- Ropinirole PR-Ropinirole PR: Participants received ropinirole PR/XR tablets orally once daily. Participants firstly received matching PR/XR placebo tablets for 2 weeks and then received 2 mg PR/XR tablets with a weekly dose increase to 4 mg at Week 4. Between Weeks 6 and 24, the dose was optionally increased at intervals of 2 weeks or longer up to 16 mg/day. In the PR/XR Switching Phase, administration of the PR/XR tablets was continued until Week 32 at the same dose level as that at the end of the Non-Inferiority Verification Phase. Participants who entered into the Long-term Phase continued to receive ropinirole PR/XR tablets until Week 54 at the same dose level as that at the end of the PR/XR Switching Phase. Participants who did not enter the Long-term Phase entered the Down-titration Phase after completion of the PR/XR Switching Phase.
- Ropinirole IR-Ropinirole PR: Participants received ropinirole IR tablets three times daily at the initial dose of 0.75 mg/day with a weekly dose increase to 3 mg/day at Week 4. Between Weeks 6 and 24, the dose was optionally increased at intervals of 2 weeks or longer up to 15 mg/day. Ropinirole IR tablets were administered until the night of the Week 24 visit and were replaced by ropinirole PR/XR tablets on the following morning, the morning of the first day of the PR/XR Switching Phase, at the same dose level. Participants who entered the Long-term Phase continued to receive ropinirole PR/XR until Week 54 at the same dose level as that at the end of the PR/XR Switching Phase. Participants who did not enter into the Long-term Phase entered the Down-titration Phase after completion of the PR/XR Switching Phase.
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 151 | 139
percentage of participants
  30 percent responder | 66 | 69
  20 percent responder | 81 | 78

3. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part I Total Score at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part I assesses mentation, behavior, and mood on 4 items. Participants receive a score of 0-4 points per item. The maximum total score is 16 points. A higher score indicates more severe mental symptoms. Mean change from Week 0 was calculated as the total score at FAP minus the total score at Week 0.
Time Frame: Week 0 and FAP (up to Week 24)
Population: FAS. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 and who had only one observation for the part I total score were not included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 151 | 142
scores on a scale | -0.2 (1.25) | -0.3 (1.21)

4. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part II (at "On") Total Score at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "On" state is defined as the state at which PD symptoms are well controlled by the drug. Mean change from Week 0 was calculated as the total score at FAP minus the score at Week 0.
Time Frame: Week 0 and FAP (up to Week 24)
Population: FAS. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 and who had only one observation for the part II (at "On") total score were not included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 151 | 142
scores on a scale | -2.6 (3.69) | -2.9 (4.17)

5. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part II (at "Off") Total Score at Week 24 in the Non-Inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Mean change from Week 0 was calculated as the total score at FAP minus the total score at Week 0. Particpants with only one observation for the part II (at "Off") total score were not included in the analysis.
Time Frame: Week 0 and FAP (up to Week 24)
Population: FAS. Only participants who had "Off" state were included in the analysis. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 were not included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 66 | 74
scores on a scale | -4.7 (4.49) | -3.8 (5.15)

6. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part IV Total Score at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part IV assesses complications of therapy on 11 items. Participants receive a score of 0-4 or 0-1 points per item depending on the item. The maximum total score is 23 points. A higher score indicates more severe symptoms of complications. Mean change from Week 0 was calculated as the total score at FAP minus the total score at Week 0.
Time Frame: Week 0 and FAP (up to Week 24)
Population: FAS. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 and who had only one observation for the part IV total score were not included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 151 | 141
scores on a scale | -0.6 (1.51) | -0.2 (1.68)

7. Secondary Outcome: Japanese UPDRS Part I Total Score at Week 0 and FAP (up to Week 24) in the Non-inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part I assesses mentation, behavior, and mood on 4 items. Participants receive a score of 0-4 points per item. The maximum total score is 16 points. A higher score indicates more severe mental symptoms.
Time Frame: Week 0 and FAP (up to Week 24)
Population: FAS. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 were not included in the analysis for the FAP.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 156 | 146
scores on a scale
  Week 0; n=156, 146 | 0.9 (1.30) | 1.1 (1.35)
  FAP; n=151, 142 | 0.7 (1.34) | 0.8 (1.50)

8. Secondary Outcome: Japanese UPDRS Part II (at "On") Total Score at Week 0 and FAP (up to Week 24) in the Non-inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "On" state is defined as the state at which PD symptoms are well controlled by the drug.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 156 | 146
scores on a scale
  Week 0; n=156, 146 | 7.7 (5.51) | 7.6 (5.87)
  FAP; n=151, 142 | 5.2 (5.21) | 4.6 (5.23)

9. Secondary Outcome: Japanese UPDRS Part II (at "Off") Total Score at Week 0 and FAP (up to Week 24) in the Non-inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug.
Time Frame: Week 0 and FAP (up to Week 24)
Population: FAS. Only participants who had "off" state were included in the analysis. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 were not included in the analysis for the FAP.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 86 | 88
scores on a scale
  Week 0; n=86, 88 | 13.6 (8.03) | 13.1 (6.64)
  FAP; n=66, 76 | 9.6 (7.24) | 8.7 (6.39)

10. Secondary Outcome: Japanese UPDRS Part III Total Score at Week 0 and FAP (up to Week 24) in the Non-inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 156 | 146
scores on a scale
  Week 0; n=156, 146 | 24.0 (9.47) | 24.3 (9.81)
  FAP; n=151, 139 | 13.7 (9.91) | 12.7 (9.39)

11. Secondary Outcome: Japanese UPDRS Part IV Total Score at Week 0 and FAP (up to Week 24) in the Non-inferiority Verification Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part IV assesses complications of therapy on 11 items. Participants receive a score of 0-4 or 0-1 points per item depending on the item. The maximum total score is 23 points. A higher score indicates more severe symptoms of complications.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 156 | 146
scores on a scale
  Week 0; n=156, 146 | 2.7 (2.59) | 2.8 (2.54)
  FAP; n=151, 141 | 2.1 (2.25) | 2.6 (2.49)

12. Secondary Outcome: Percentage of Responders on the Clinical Global Impression-Improvement (CGI-I) at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: The CGI-I assesses the participant's improvement or worsening of PD from Baseline with the following eight grades: 0 = Not Assessed, 1 = Very Much Improved, 2 = Much Improved, 3 = Minimally Improved, 4 = No Change, 5 = Minimally Worse, 6 = Much Worse, and 7 = Very Much Worse. Responders are defined as those participants with scores of very much improved or much improved.
Time Frame: FAP (up to Week 24)
Population: FAS. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 151 | 142
percentage of participants | 63 | 61

13. Secondary Outcome: Percentage of Responders in Change From Week 0 in Awake Time Spent "Off" at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Responders were defined as participants with a 20 percent or greater reduction on change from Week 0 in Off time (percentage).
Time Frame: FAP (up to Week 24)
Population: FAS. Participants who had 0 hour as Off time at Week 0 were excluded from the analysis. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 78 | 77
percentage of participants | 44 | 40

14. Secondary Outcome: Percentage of Responders in Percent Change From Week 0 in Awake Time Spent "Off" at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Responders were defined as participants with a 20 percent or greater reduction in percent change from Week 0 in Off time (percentage).
Time Frame: FAP (up to Week 24)
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 78 | 77
percentage of participants | 76 | 69

15. Secondary Outcome: Mean Change From Week 0 in Awake Time Spent "Off" at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Mean change from Week 0 in Off time (actual hours) was calculated as Off time (hours) at FAP minus Off time (hours) at Week 0.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 78 | 77
hours | -2.88 (3.941) | -2.59 (4.691)

16. Secondary Outcome: Mean Change From Week 0 in Percentage of Awake Time Spent "Off" at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. "Off" time is measured as a proportion using the following formula: (Sum of two days off time [hours]/Sum of two days awake time [hours]) x 100. Change from Week 0 in Off time is measured using the following formula: Off time (proportion) at FAP minus Off time (proportion) at Week 0.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 78 | 77
percentage of time | -18.39 (23.600) | -16.81 (27.150)

17. Secondary Outcome: Mean Percent Change From Week 0 in Percentage of Awake Time Spent "Off" at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. "Off" time is measured as a proportion using the following formula: (Sum of two days off time [hours]/Sum of two days awake time [hours]) x 100. Percent change from Week 0 in Off time (proportion) is measured using the following formula: (Change from Week 0 in Off time [proportion]/Off time [proportion] at Week 0) x 100.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 78 | 77
percent change | -42.36 (77.250) | -40.48 (60.344)

18. Secondary Outcome: Mean Change From Week 0 in Awake Time Spent "On" at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Mean Change from Week 0 in On time (actual hours) was calculated as On time (hours) at FAP minus On time (hours) at Week 0. Participants who had only one observation for On time were not included in the analysis.
Time Frame: Week 0 and FAP (up to Week 24)
Population: FAS. Participants who had 0 hour as On time at Week 0 were excluded from the analysis. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 were not included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 149 | 134
hours | 1.65 (3.215) | 1.35 (3.539)

19. Secondary Outcome: Mean Change From Week 0 in Percentage of Awake Time Spent "On" at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. "On" time is measured as a proportion using the following formula: (Sum of two days On time [hours]/Sum of two days awake time [hours]) x 100. Change from Week 0 in On time is measured using the following formula: On time (proportion) at FAP minus On time (proportion) at Week 0. Participants who had only one observation for On time were not included in the analysis.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 149 | 134
percentage of time | 9.03 (18.634) | 7.79 (19.895)

20. Secondary Outcome: Mean Change From Week 0 in Awake Time Spent "On" With Troublesome Dyskinesias at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Troublesome dyskinesia is defined as dyskinesia that interferes with the participant's daily activity. Mean change from Week 0 in On time with troublesome dyskinesias (actual hours) was calculated as On time with troublesome dyskinesias (hours) at FAP minus On time with troublesome dyskinesias (hours) at Week 0. Participants who had only one observation for On time with troublesome dyskinesias were not included in the analysis.
Time Frame: Week 0 and FAP (up to Week 24)
Population: FAS. Participants who had 0 hour as On time with troublesome dyskinesias at Week 0 were excluded from the analysis. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include values of Weeks 0, 1, and 2; participants who withdrew before Week 2 were not included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 7 | 13
hours | 0.57 (3.886) | 0.87 (2.311)

21. Secondary Outcome: Mean Change From Week 0 in Percentage of Awake Time Spent "On" With Troublesome Dyskinesias at FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: "On" time with troublesome dyskinesias is measured as a proportion using the following formula: (Sum of two days On time with troublesome dyskinesias [hours]/Sum of two days awake time [hours]) x 100. Change from Week 0 in On time with troublesome dyskinesias is measured using the following formula: On time with troublesome dyskinesias (proportion) at FAP minus On time with troublesome dyskinesias (proportion) at Week 0. Participants who had only one observation for On time with troublesome dyskinesias were not included in the analysis.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 2 | 13
percentage of time | 2.61 (24.247) | 5.39 (14.399)

22. Secondary Outcome: Number of Participants at Each Stage of the Modified Hoehn & Yahr Severity of Illness (at "On") at Week 0 and FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: The Modified Hoehn & Yahr criteria are measured on the following 8-point scale for disease severity: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease; 2.5, Mild bilateral disease; 3, Mild to moderate bilateral disease; 4, Severe disability; and 5, Wheelchair bound or bedridden unless aided. "On" state is defined as the state at which PD symptoms are well controlled by the drug.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 156 | 146
participants
  Week 0; Stage 0; n=156, 146 | 0 | 0
  Week 0; Stage 1; n=156, 146 | 0 | 0
  Week 0; Stage 1.5; n=156, 146 | 0 | 1
  Week 0; Stage 2; n=156, 146 | 34 | 34
  Week 0; Stage 2.5; n=156, 146 | 47 | 43
  Week 0; Stage 3; n=156, 146 | 64 | 57
  Week 0; Stage 4; n=156, 146 | 11 | 10
  Week 0; Stage 5; n=156, 146 | 0 | 1
  FAP; Stage 0; n=151, 142 | 2 | 4
  FAP; Stage 1; n=151, 142 | 20 | 18
  FAP; Stage 1.5; n=151, 142 | 3 | 14
  FAP; Stage 2; n=151, 142 | 54 | 44
  FAP; Stage 2.5; n=151, 142 | 31 | 29
  FAP; Stage 3; n=151, 142 | 34 | 27
  FAP; Stage 4; n=151, 142 | 7 | 6
  FAP; Stage 5; n=151, 142 | 9 | 0

23. Secondary Outcome: Number of Participants at Each Stage of the Modified Hoehn & Yahr Severity of Illness (at "Off") at Week 0 and FAP (up to Week 24) in the Non-Inferiority Verification Phase
Description: The Modified Hoehn & Yahr criteria are measured on the following 8-point scale for disease severity: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease; 2.5, Mild bilateral disease; 3, Mild to moderate bilateral disease; 4, Severe disability; and 5, Wheelchair bound or bedridden unless aided. "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug.
Time Frame: Week 0 and FAP (up to Week 24)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 86 | 88
participants
  Week 0; Stage 0; n=86, 88 | 0 | 0
  Week 0; Stage 1; n=86, 88 | 0 | 0
  Week 0; Stage 1.5; n=86, 88 | 0 | 0
  Week 0; Stage 2; n=86, 88 | 4 | 7
  Week 0; Stage 2.5; n=86, 88 | 13 | 14
  Week 0; Stage 3; n=86, 88 | 39 | 37
  Week 0; Stage 4; n=86, 88 | 24 | 26
  Week 0; Stage 5; n=86, 88 | 6 | 4
  FAP; Stage 0; n=66, 76 | 0 | 0
  FAP; Stage 1; n=66, 76 | 5 | 2
  FAP; Stage 1.5; n=66, 76 | 3 | 1
  FAP; Stage 2; n=66, 76 | 9 | 23
  FAP; Stage 2.5; n=66, 76 | 13 | 11
  FAP; Stage 3; n=66, 76 | 19 | 22
  FAP; Stage 4; n=66, 76 | 15 | 14
  FAP; Stage 5; n=66, 76 | 2 | 3

24. Secondary Outcome: Percentage of Participants Remaining in the Study on the Indicated Days During the Non-Inferiority Verification Phase in the Ropinirole PR-Ropinirole PR Group
Description: The percentage of participants remaining in the study was presented by Kaplan-Meier method, where premature discontinuation (i.e., withdrawal before Week 24) was the event, and participants who had completed the phase were censored.
Time Frame: 0-175 days (up to Week 24)
Population: FAS. Data were evaluated only at the time point at which they had been collected.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 156
percentage of participants
  0 days | 100
  6 days | 99
  9 days | 99
  14 days | 98
  17 days | 97
  19 days | 96
  20 days | 96
  21 days | 93
  25 days | 92
  28 days | 91
  34 days | 90
  42 days | 90
  43 days | 89
  55 days | 88
  62 days | 88
  74 days | 87
  119 days | 86
  139 days | 85
  142 days | 85
  153 days | 84
  154 days | 83
  160 days | 83
  168 days | 82
  175 days | 82

25. Secondary Outcome: Percentage of Participants Remaining in the Study on the Indicated Days During the Non-Inferiority Verification Phase in the Ropinirole IR-Ropinirole PR Group
Description: as for outcome 24
Time Frame: 0-175 days (up to Week 24)
Population: FAS. Data were evaluated only at the time point at which they had been collected.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 146
percentage of participants
  0 days | 100
  7 days | 99
  12 days | 99
  14 days | 97
  18 days | 97
  21 days | 96
  28 days | 94
  30 days | 93
  32 days | 92
  42 days | 90
  51 days | 90
  55 days | 88
  60 days | 88
  86 days | 87
  88 days | 86
  119 days | 86
  142 days | 85
  168 days | 84
  175 days | 84

26. Secondary Outcome: Mean Change From Week 24 (Period Baseline) in the Japanese UPDRS Part I Total Score at FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part I assesses mentation, behavior, and mood on 4 items. Participants receive a score of 0-4 points per item. The maximum total score is 16 points. A higher score indicates more severe mental symptoms. Mean change from Week 24 was calculated as the total score at FAP minus the total score at Week 24. Participants whose observation could not be obtained after Week 24 because of their premature withdrawal or other reasons were not included.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: Switching-FAS: participants who were included in the FAS and progressed to the PR/XR Switching Phase. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include Week 24 values.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 127 | 120
scores on a scale | -0.0 (0.40) | 0.1 (0.45)

27. Secondary Outcome: Mean Change From Week 24 in the Japanese UPDRS Part II (at "On") Total Score at FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "On" state is defined as the state at which PD symptoms are well controlled by the drug. Mean change from Week 24 was calculated as the total score at FAP minus the total score at Week 24.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: Switching-FAS. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include Week 24 values. Participants whose observation could not be obtained after Week 24 because of their premature withdrawal or other reasons were not included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 126 | 119
scores on a scale | -0.0 (1.37) | 0.3 (1.77)

28. Secondary Outcome: Mean Change From Week 24 in the Japanese UPDRS Part II (at "Off") Total Score at FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "Off" state is where PD symptoms are not adequately controlled by the drug. Mean change from Week 0 was calculated as the total score at FAP minus the total score at Week 0. Participants whose observation could not be obtained after Week 24 because of their premature withdrawal or other reasons were not included in the analysis.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: Switching-FAS. Only participants who had "off" state were included in the analysis. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include Week 24 values.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 57 | 60
scores on a scale | -0.2 (1.89) | -0.4 (2.35)

29. Secondary Outcome: Mean Change From Week 24 in the Japanese UPDRS Part III Total Score at FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. Mean change from Week 24 was calculated as the total score at FAP minus the total score at Week 24.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 125 | 117
scores on a scale | -0.2 (2.81) | -0.7 (3.17)

30. Secondary Outcome: Mean Change From Week 24 in the Japanese UPDRS Part IV Total Score at FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part IV assesses complications of therapy on 11 items. Participants receive a score of 0-4 or 0-1 points per item depending on the item. The maximum total score is 23 points. A higher score indicates more severe symptoms of complications. Mean change from Week 24 was calculated as the total score at FAP minus the total score at Week 24.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 127 | 119
scores on a scale | -0.1 (0.64) | -0.2 (1.04)

31. Secondary Outcome: Japanese UPDRS Part I Total Score at Week 24 and FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: as for outcome 7
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: Switching-FAS. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include Week 24 values. Participants whose observation could not be obtained after Week 24 because of their premature withdrawal or other reasons were not included in the analysis for the FAP.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 127 | 122
scores on a scale
  Week 24; n=127, 122 | 0.5 (0.96) | 0.6 (1.22)
  FAP; n=127, 120 | 0.4 (1.04) | 0.7 (1.34)

32. Secondary Outcome: Japanese UPDRS Part II (at "On") Total Score at Week 24 and FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: as for outcome 8
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 127 | 122
scores on a scale
  Week 24; n=127, 122 | 4.4 (4.59) | 4.1 (4.60)
  FAP; n=126, 119 | 4.4 (4.59) | 4.3 (4.88)

33. Secondary Outcome: Japanese UPDRS Part II (at "Off") Total Score at Week 24 and FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Only participants who had "off" state were included in the analysis.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 58 | 63
scores on a scale
  Week 24; n=58, 63 | 8.8 (6.80) | 7.8 (5.57)
  FAP; n=57, 61 | 8.5 (7.31) | 7.5 (5.78)

34. Secondary Outcome: Japanese UPDRS Part III Total Score at Week 24 and FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. One participant whose observation could not be obtained at Week 24 was not included in the analysis for Week 24.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 127 | 121
scores on a scale
  Week 24; n=127, 121 | 11.9 (8.63) | 12.3 (8.91)
  FAP; n=125, 118 | 11.7 (8.23) | 11.3 (8.86)

35. Secondary Outcome: Japanese UPDRS Part IV Total Score at Week 24 and FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part IV assesses complications of therapy on 11 items. Participants receive a score of 0-4 or 0-1 points per item depending on the item. The maximum total score is 23 points. A higher score indicates more severe symptoms of complications. One participant whose observation could not be obtained at Week 24 was not included in the analysis for Week 24.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 127 | 121
scores on a scale
  Week 24; n=127, 121 | 1.9 (2.14) | 2.5 (2.47)
  FAP; n=127, 119 | 1.9 (2.17) | 2.3 (2.32)

36. Secondary Outcome: Mean Change From Week 24 in Awake Time Spent "Off" at FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Mean change from Week 24 in Off time (actual hours) was calculated as Off time (hours) at FAP minus Off time (hours) at Week 24. Participants whose observation could not be obtained after Week 24 because of their premature withdrawal or other reasons were not included in the analysis.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: Switching-FAS. Participants who had 0 hour as Off time at Week 24 were excluded from the analysis. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include Week 24 values.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 51 | 52
hours | -0.07 (2.912) | -0.13 (2.005)

37. Secondary Outcome: Mean Change From Week 24 in Percentage of Awake Time Spent "Off" at FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. "Off" time is measured as a proportion using the following formula: (Sum of two days off time [hours]/Sum of two days awake time [hours]) x 100. Change from Week 24 in Off time is measured using the following formula: Off time (proportion) at FAP minus Off time (proportion) at Week 24. Participants whose observation could not be obtained after Week 24 because of their premature withdrawal or other reasons were not included in the analysis.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 51 | 52
percentage of time | -0.97 (16.470) | -0.14 (12.913)

38. Secondary Outcome: Mean Change From Week 24 in Awake Time Spent "On" With Troublesome Dyskinesias at FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Troublesome dyskinesia is defined as dyskinesia that interferes with the participant's daily activity. Mean change from Week 24 on On time with troublesome dyskinesias (actual hours) was calculated as On time with troublesome dyskinesias (hours) at FAP minus On time with troublesome dyskinesias (hours) at Week 24. Participants who had 0 hour as On time with troublesome dyskinesias at Week 24 were excluded from the analysis.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: Switching-FAS. On-treatment last observations within the phase were carried forward as FAP values of the phase. FAP values do not include Week 24 values. Participants whose observation could not be obtained after Week 24 because of their premature withdrawal or other reasons were also not included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 9 | 12
hours | 0.00 (3.180) | -1.25 (1.831)

39. Secondary Outcome: Number of Participants at Each Stage of the Modified Hoehn & Yahr Severity of Illness (at "On") at Week 24 and FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: as for outcome 22
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 31
Measure: Number; unit: participants
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 127 | 122
participants
  Week 24; Stage 0; n=127, 122 | 2 | 4
  Week 24; Stage 1; n=127, 122 | 20 | 16
  Week 24; Stage 1.5; n=127, 122 | 3 | 12
  Week 24; Stage 2; n=127, 122 | 49 | 41
  Week 24; Stage 2.5; n=127,122 | 25 | 24
  Week 24; Stage 3; n=127, 122 | 22 | 23
  Week 24; Stage 4; n=127, 122 | 6 | 2
  Week 24; Stage 5; n=127, 122 | 0 | 0
  FAP; Stage 0; n=125, 119 | 3 | 3
  FAP; Stage 1; n=125, 119 | 17 | 19
  FAP; Stage 1.5; n=125, 119 | 5 | 10
  FAP; Stage 2; n=125, 119 | 51 | 44
  FAP; Stage 2.5; n=125, 119 | 23 | 20
  FAP; Stage 3; n=125, 119 | 20 | 20
  FAP; Stage 4; n=125, 119 | 6 | 2
  FAP; Stage 5; n=125, 119 | 0 | 1

40. Secondary Outcome: Number of Participants at Each Stage of the Modified Hoehn & Yahr Severity of Illness (at "Off") at Week 24 and FAP (From Week 26 up to Week 32) in the PR/XR Switching Phase
Description: The Modified Hoehn & Yahr criteria are measured on the following 8-point scale for disease severity: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease; 2.5, Mild bilateral disease; 3, Mild to moderate bilateral disease; 4, Severe disability; and 5, Wheelchair bound or bedridden unless aided. "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Only participants who had "off" state were included in the analysis.
Time Frame: Week 24 and FAP (from Week 26 up to Week 32)
Population: as for outcome 31
Measure: Number; unit: participants
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 58 | 63
participants
  Week 24; Stage 0; n=58, 63 | 0 | 0
  Week 24; Stage 1; n=58, 63 | 5 | 2
  Week 24; Stage 1.5; n=58, 63 | 3 | 0
  Week 24; Stage 2; n=58, 63 | 9 | 21
  Week 24; Stage 2.5; n=58, 63 | 13 | 11
  Week 24; Stage 3; n=58, 63 | 14 | 18
  Week 24; Stage 4; n=58, 63 | 13 | 9
  Week 24; Stage 5; n=58, 63 | 1 | 2
  FAP; Stage 0; n=56, 61 | 0 | 0
  FAP; Stage 1; n=56, 61 | 4 | 3
  FAP; Stage 1.5; n=56, 61 | 3 | 0
  FAP; Stage 2; n=56, 61 | 12 | 16
  FAP; Stage 2.5; n=56, 61 | 13 | 15
  FAP; Stage 3; n=56, 61 | 11 | 18
  FAP; Stage 4; n=56, 61 | 11 | 7
  FAP; Stage 5; n=56, 61 | 2 | 2

41. Secondary Outcome: Percentage of Participants Remaining in the Study on the Indicated Days During the PR/XR Switching Phase in the Ropinirole PR-Ropinirole PR Group
Description: The percentage of participants remaining in the study was presented by Kaplan-Meier method, where premature discontinuation (i.e., withdrawal before Week 32) was the event, and participants who had completed the phase were censored.
Time Frame: 0-89 days within the PR/XR Switching Phase (between Weeks 24 and 32)
Population: Switching-FAS. Data were evaluated only at the time point at which they had been collected.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 127
percentage of participants
  0 days | 100
  28 days | 99
  35 days | 98
  89 days | 98

42. Secondary Outcome: Percentage of Participants Remaining in the Study on the Indicated Days During the PR/XR Switching Phase in the Ropinirole IR-Ropinirole PR Group
Description: as for outcome 41
Time Frame: 0-89 days within the PR/XR Switching Phase (between Weeks 24 and 32)
Population: Switching-FAS. Data were evaluated only at the time point at which they had been collected.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole IR-Ropinirole PR
Number analyzed (Participants) | 122
percentage of participants
  0 days | 100
  4 days | 99
  7 days | 98
  18 days | 98
  28 days | 97
  33 days | 96
  89 days | 96

43. Secondary Outcome: Percentage of Responders on the Japanese UPDRS Part III Total Score at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: Thirty percent responders were defined as participants with a 30 percent or greater reduction from Week 0 (Baseline) in the Japanese UPDRS Part III total score. Twenty percent responders were defined as participants with a 20 percent or greater reduction from Week 0 in the Japanese UPDRS Part III total score.
Time Frame: Week 54
Population: Long-FAS: participants who were included in the FAS and entered into the Long-term Phase. Data were evaluated only at the time point at which they had been collected; participants whose observation could not be obtained because of their premature withdrawal or other reasons were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 68
percentage of participants
  30 percent responders | 84
  20 percent responders | 76

44. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part I Total Score at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part I assesses mentation, behavior, and mood on 4 items. Participants receive a score of 0-4 points per item. The maximum total score is 16 points. A higher score indicates more severe mental symptoms. Mean change from Week 0 was calculated as the total score at Week 54 minus the total score at Week 0.
Time Frame: Weeks 0 and 54
Population: Long-FAS. Data were evaluated only at the time point at which they had been collected; participants whose observation could not be obtained because of their premature withdrawal or other reasons were not included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 68
scores on a scale | -0.4 (0.95)

45. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part II (at "On") Total Score at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "On" state is defined as the state at which PD symptoms are well controlled by the drug. Mean change from Week 0 was calculated as the total score at Week 54 minus the total score at Week 0.
Time Frame: Weeks 0 and 54
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 67
scores on a scale | -2.6 (4.23)

46. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part II (at "Off") Total Score at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part II assesses activities of daily living on 13 items. Participants receive a score of 0-4 points per item. The maximum total score is 52 points. A higher score indicates more severe PD symptoms. "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Mean change from Week 0 was calculated as the total score at Week 54 minus the total score at Week 0.
Time Frame: Weeks 0 and 54
Population: Long-FAS. Only participants who had "off" state were included in the analysis. Data were evaluated only at the time point at which they had been collected; participants whose observation could not be obtained because of their premature withdrawal or other reasons were not included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 32
scores on a scale | -4.6 (3.83)

47. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part III Total Score at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part III assesses motor examination on 27 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. Mean change from Week 0 was calculated as the total score at Week 54 minus the total score at Week 0.
Time Frame: Weeks 0 and 54
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 68
scores on a scale | -12.7 (8.23)

48. Secondary Outcome: Mean Change From Week 0 in the Japanese UPDRS Part IV Total Score at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: The Japanese UPDRS assesses the status of PD patients objectively. Part IV assesses complications of therapy on 11 items. Participants receive a score of 0-4 or 0-1 points per item depending on the item. The maximum total score is 23 points. A higher score indicates more severe symptoms of complications. Mean change from Week 0 was calculated as the total score at Week 54 minus the total score at Week 0.
Time Frame: Weeks 0 and 54
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 68
scores on a scale | -0.8 (1.52)

49. Secondary Outcome: Japanese UPDRS Part I Total Score at Weeks 0 and 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: as for outcome 7
Time Frame: Weeks 0 and 54
Population: Long-FAS. Data were evaluated only at the time point at which they had been collected; participants whose observation could not be obtained because of their premature withdrawal or other reasons were not included in the analysis for Week 54.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 73
scores on a scale
  Week 0, n=73 | 1.1 (1.34)
  Week 54, n=68 | 0.6 (0.93)

50. Secondary Outcome: Japanese UPDRS Part II (at "On") Total Score at Weeks 0 and 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: as for outcome 8
Time Frame: Weeks 0 and 54
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 73
scores on a scale
  Week 0, n=73 | 6.9 (4.57)
  Week 54, n=67 | 4.3 (4.38)

51. Secondary Outcome: Japanese UPDRS Part II (at "Off") Total Score at Weeks 0 and 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: as for outcome 9
Time Frame: Weeks 0 and 54
Population: Long-FAS. Only participants who had "off" state were included in the analysis. Data were evaluated only at the time point at which they had been collected; participants whose observation could not be obtained because of their premature withdrawal or other reasons were not included in the analysis for Week 54.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 44
scores on a scale
  Week 0, n=44 | 13.2 (7.40)
  Week 54, n=32 | 9.0 (6.74)

52. Secondary Outcome: Japanese UPDRS Part III Total Score at Weeks 0 and 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: as for outcome 10
Time Frame: Weeks 0 and 54
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 73
scores on a scale
  Week 0, n=73 | 24.6 (8.54)
  Week 54, n=68 | 11.9 (8.08)

53. Secondary Outcome: Japanese UPDRS Part IV Total Score at Weeks 0 and 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: as for outcome 11
Time Frame: Weeks 0 and 54
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 73
scores on a scale
  Week 0, n=73 | 2.9 (2.69)
  Week 54, n=68 | 2.1 (2.28)

54. Secondary Outcome: Percentage of Responders on the CGI-I at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: as for outcome 12
Time Frame: Week 54
Population: as for outcome 44
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 68
percentage of participants | 65

55. Secondary Outcome: Percentage of Responders in Change From Week 0 in Awake Time Spent "Off" at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Responders were defined as participants with a 20 percent or greater reduction in change from Week 0 in Off time (percentage).
Time Frame: Week 54
Population: Long-FAS. Participants who had 0 hour as Off time at Week 0 were excluded from the analysis. Data were evaluated only at the time point at which they had been collected; participants whose observation could not be obtained because of their premature withdrawal or other reasons were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 39
percentage of participants | 46

56. Secondary Outcome: Percentage of Responders in Percent Change From Week 0 in Awake Time Spent "Off" at Week 54 in the Long-term Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Responders were defined as participants with a 20 percent or greater reduction on percent change from Week 0 in Off time (percentage).
Time Frame: Week 54
Population: as for outcome 55
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 39
percentage of participants | 79

57. Secondary Outcome: Mean Change From Week 0 in Awake Time Spent "Off" at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Mean change from Week 0 in Off time (actual hours) was calculated as Off time (hours) at Week 54 minus Off time (hours) at Week 0.
Time Frame: Weeks 0 and 54
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 39
hours | -2.87 (3.642)

58. Secondary Outcome: Mean Change From Week 0 in Percentage of Awake Time Spent "Off" at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. "Off" time is measured as a proportion using the following formula: (Sum of two days off time [hours]/Sum of two days awake time [hours]) x 100. Change from Week 0 in Off time is measured using the following formula: Off time (proportion) at Week 54 minus Off time (proportion) at Week 0.
Time Frame: Weeks 0 and 54
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 39
percentage of time | -18.55 (23.038)

59. Secondary Outcome: Mean Change From Week 0 in Awake Time Spent "On" With Troublesome Dyskinesias at Week 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Troublesome dyskinesia is defined as dyskinesia that interferes with the participant's daily activity. Mean change from Week 0 in On time with troublesome dyskinesias (actual hours) was calculated as On time with troublesome dyskinesias (hours) at Week 54 minus On time with troublesome dyskinesias (hours) at Week 0.
Time Frame: Weeks 0 and 54
Population: Long-FAS. Participants who had 0 hour as On time with troublesome dyskinesias at Week 0 were excluded from the analysis. Data were evaluated only at the time point at which they had been collected; participants whose observation could not be obtained because of their premature withdrawal or other reasons were not included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 3
hours | -0.33 (0.629)

60. Secondary Outcome: Number of Participants at Each Stage of the Modified Hoehn & Yahr Severity of Illness (at "On") at Weeks 0 and 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: as for outcome 22
Time Frame: Weeks 0 and 54
Population: as for outcome 49
Measure: Number; unit: participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 73
participants
  Week 0; Stage 0; n=73 | 0
  Week 0; Stage 1; n=73 | 0
  Week 0; Stage 1.5; n=73 | 0
  Week 0; Stage 2; n=73 | 18
  Week 0; Stage 2.5; n=73 | 19
  Week 0; Stage 3; n=73 | 35
  Week 0; Stage 4; n=73 | 1
  Week 0; Stage 5; n=73 | 0
  Week 54; Stage 0; n=67 | 1
  Week 54; Stage 1; n=67 | 8
  Week 54; Stage 1.5; n=67 | 3
  Week 54; Stage 2; n=67 | 29
  Week 54; Stage 2.5; n=67 | 15
  Week 54; Stage 3; n=67 | 11
  Week 54; Stage 4; n=67 | 0
  Week 54; Stage 5; n=67 | 0

61. Secondary Outcome: Number of Participants at Each Stage of the Modified Hoehn & Yahr Severity of Illness (at "Off") at Weeks 0 and 54 in the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: as for outcome 23
Time Frame: Weeks 0 and 54
Population: as for outcome 51
Measure: Number; unit: participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 44
participants
  Week 0; Stage 0; n=44 | 0
  Week 0; Stage 1; n=44 | 0
  Week 0; Stage 1.5; n=44 | 0
  Week 0; Stage 2; n=44 | 2
  Week 0; Stage 2.5; n=44 | 8
  Week 0; Stage 3; n=44 | 21
  Week 0; Stage 4; n=44 | 11
  Week 0; Stage 5; n=44 | 2
  Week 54; Stage 0; n=32 | 0
  Week 54; Stage 1; n=32 | 3
  Week 54; Stage 1.5; n=32 | 1
  Week 54; Stage 2; n=32 | 5
  Week 54; Stage 2.5; n=32 | 9
  Week 54; Stage 3; n=32 | 6
  Week 54; Stage 4; n=32 | 7
  Week 54; Stage 5; n=32 | 1

62. Secondary Outcome: Percentage of Participants Remaining in the Study on the Indicated Days During the Long-term Phase in the Ropinirole PR-Ropinirole PR Group
Description: The percentage of participants remaining in the study was presented by Kaplan-Meier method, where premature discontinuation (i.e., withdrawal before Week 54) was the event, and participants who had completed the study were censored.
Time Frame: 0-385 days (up to Week 54)
Population: Long-FAS. Data were evaluated only at the time point at which they had been collected.
Measure: Number; unit: percentage of participants
Arm/Group | Ropinirole PR-Ropinirole PR
Number analyzed (Participants) | 73
percentage of participants
  0 days | 100
  258 days | 99
  261 days | 97
  322 days | 96
  329 days | 95
  346 days | 93
  385 days | 93

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the start of investigational product until follow-up contact (up to 61 weeks). Other (non-serious) adverse events were collected from Baseline through Week 54.
Description: Baseline for other (non-serious) adverse events: Week 2 for ropinirole PR-ropinirole PR group, Week 0 for ropinirole IR-ropinirole PR group
Arm/Group | Ropinirole PR-Ropinirole PR | Ropinirole IR-Ropinirole PR
Serious Adverse Events (participants affected / at risk) | 16/156 | 16/146
Other Adverse Events (participants affected / at risk) | 95/156 | 98/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole PR-Ropinirole PR (N=156) | Ropinirole IR-Ropinirole PR (N=146)
Cerebral infarction (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood pressure orthostatic decreased (Investigations) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole PR-Ropinirole PR (N=156) | Ropinirole IR-Ropinirole PR (N=146)
Somnolence (Nervous system disorders) | 18 | 17
Dyskinesia (Nervous system disorders) | 9 | 17
Dizziness (Nervous system disorders) | 3 | 12
Nausea (Gastrointestinal disorders) | 20 | 17
Constipation (Gastrointestinal disorders) | 14 | 11
Vomiting (Gastrointestinal disorders) | 9 | 5
Nasopharyngitis (Infections and infestations) | 30 | 29
Hallucination (Psychiatric disorders) | 14 | 9
Insomnia (Psychiatric disorders) | 4 | 8
Contusion (Injury, poisoning and procedural complications) | 9 | 7
Fall (Injury, poisoning and procedural complications) | 9 | 6
Orthostatic hypotension (Vascular disorders) | 10 | 11
Decreased appetite (Metabolism and nutrition disorders) | 11 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.